CLINICAL TRIAL: NCT03274635
Title: Desk-Compatible Elliptical Device: Feasibility Evaluation
Brief Title: Penn State Hershey Sitting and Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Liza Rovniak, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21HL118453 (NIH)
Record Dates: First submitted 2017-09-01; First posted 2017-09-07 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Usual Delayed Compensation, Money (Active Comparator): Will receive delayed monetary compensation with Amazon gift card, non performance-contingent.
  Interventions: Behavioral: Desk-based pedaling device and pedaling incentives provided
- Usual Delayed Compensation, Food (Active Comparator): Will receive delayed compensation with food-based gift card, non performance-contingent.
  Interventions: Behavioral: Desk-based pedaling device and pedaling incentives provided
- Individual Immediate Contingent Reward, Money (Experimental): Will receive daily performance-contingent monetary compensation with Amazon gift card.
  Interventions: Behavioral: Desk-based pedaling device and pedaling incentives provided
- Individual Immediate Contingent Reward, Food (Experimental): Will receive daily performance-contingent food-based gift card.
  Interventions: Behavioral: Desk-based pedaling device and pedaling incentives provided
- Joint Immediate Contingent Reward, Money (Experimental): Will receive daily performance-contingent monetary compensation with Amazon gift card, with additional compensation contingent on pedaling activity of co-worker participant.
  Interventions: Behavioral: Desk-based pedaling device and pedaling incentives provided
- Joint Immediate Contingent Reward, Food (Experimental): Will receive daily performance-contingent monetary compensation with food gift card, with additional compensation contingent on pedaling activity of co-worker participant.
  Interventions: Behavioral: Desk-based pedaling device and pedaling incentives provided

INTERVENTIONS:
Behavioral: Desk-based pedaling device and pedaling incentives provided — Varying types of incentives, equivalent in monetary value, will be randomly assigned across the 6 arms to promote regular desk-based pedaling. A free desk-based pedaling device will be provided. Effects on amount of desk-based pedaling and work productivity will be evaluated.

SUMMARY:
The purpose of this study is to: (a) evaluate if a desk-based elliptical device can help employees to increase their daily physical activity without compromising work productivity; and (b) evaluate the effects of different types of incentives for pedaling the desk-based elliptical device on employees' pedaling quantity over a one-month intervention period. The study will involve placing a compact elliptical device (provided at no cost by the research team) under employees' desk at Penn State Hershey Medical Center/College of Medicine. Data evaluating the effects of the elliptical device on work productivity will be obtained from both employees and the employees' supervisors.

ELIGIBILITY:
Inclusion Criteria:

* Full time employee, employed at least 35 hours per week at Penn State Hershey
* Able to provide documented approval from supervisor to participate
* Age 18-70 years
* Overweight or obese (BMI between 25-55)
* Sit at desk at least 5 hours per day
* Have regular working hours between 6 am and 6 pm on weekdays
* Ability to understand written and spoken English
* Own a smartphone (Android or iPhone) with Internet access
* Willing to download cycling app on smartphone during one month study period

Exclusion Criteria:

* Not present in Penn State Hershey office during study period due to personal circumstances such as travel/extended vacation or leave, relocation, or health-related circumstances
* Advised to only do physical activity recommended by a physician
* Chest pain during physical activity or during prior month
* Currently has a desk-based pedaling device or treadmill workstation already installed at desk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Change in Worker Productivity | Baseline (1 month period prior to program start) and post-program (immediately after program ends)
  Self-report assessments of worker productivity. The assessments will ask about work productivity in the prior 4-week period.
Elliptical Device Pedaling Quantity | 1 month (4 weeks) during pedaling program
  Objectively-measured pedaling quantity from elliptical device

SECONDARY OUTCOMES:
User satisfaction, process evaluations | Post-program (immediately after program ends)
  Satisfaction with intervention condition
General (non-desk pedaling) physical activity | Baseline (1 month period prior to program start) and post-program (immediately after program ends)
  Self-reported physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No